CLINICAL TRIAL: NCT02038751
Title: The Phenotyping and Genotyping of Taiwanese Patients With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201306007RINB
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Genotyping; Phenotyping; Sleep Apnea; Genetic Association Studies; Phenotype
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Index proband: moderate to severe OSA (AHI>30 or AHI>15 needing CPAP intervention) age 20-99 y/o
- Index family: first-degree, second-degree, or spouse of index proband age >20 y/o
- Control proband: friends of index proband, living in the same environment as index proband age > 20 y/o
- Control family: first-degree, second-degree, or spouse of control proband age >20 y/o

SUMMARY:
The growing evidence showed that the OSA is a heritable complex genetic disease where the genetic basis contributed the development of OSA and its sequel. The phenotyping of OSA include high level and intermediate level. The former indicates the AHI, and later includes craniofacial morphology, ventilator control, obesity, and sleepiness vulnerability.

Many studies tried to determine the association of candidate genes with OSA through association studies. However, the results were conflicting. We identified 37 candidate genes involved in six biologic pathways of OSA reported in previous literatures, including oxidative phosphorylation, cell signaling, apoptosis, cellular adhesion and motility, cell cycle, and cytokine/chemokine.

To investigate the association between phenotype and genotype of OSA, we conducted this cross-sectional study by recruiting the patients of moderate-severe OSA (index proband) and their first and second-degree family members, and friends and their family members (control family) and using candidate genes reported in the literature and whole genome SNP array for genotype approach.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized with recurrent collapse of upper airway during sleep resulting in hypoxia and sleep fragmentation. Patients of OSA might have symptoms like snoring, non-restorative sleep, witnessed apnea, and excessive daytime sleepiness. Currently, polysomnography is the gold standard for diagnosing OSA and the apnea-hypopnea index (AHI) is the parameters to indicate the severity of OSA. However, AHI poorly correlated with clinical severity of OSA, where the symptoms of patients with the identical AHI could vary from minimal to striking. The sequels of OSA include cardiovascular diseases, metabolic disorders, and neurocognitive dysfunctions. Till now, continuous positive airway pressure (CPAP) is the standard treatment for OSA where it can effectively improve daytime sleepiness, blood pressure, metabolic abnormalities, and quality of life, especially in patients with daytime sleepiness.

The growing evidence showed that the OSA is a heritable complex genetic disease where the genetic basis contributed the development of OSA and its sequel. The phenotyping of OSA include high level and intermediate level. The former indicates the AHI, and later includes craniofacial morphology, ventilator control, obesity, and sleepiness vulnerability. Many studies tried to determine the association of candidate genes with OSA through association studies. However, the results were conflicting. To clarify the influence of genotyping on phenotyping, we reported a Chinese family with congenital central hypoventilation syndrome (CCHS) that had a clinical spectrum ranging from newborn fatality to adulthood. Genetic analysis was used to confirm the presence of the PHOX2B expansion mutation. Moreover, to clarify the association between ACE I/D polymorphisms and OSA, we undertook a meta-analysis on all studies published in this area. It has not demonstrated an association between the ACE I/D polymorphism and OSA susceptibility irrespective of ethnicity, population sample or the presence/absence of co-morbid hypertension.

Nowadays, a couple of studies tried to genome-wide profiled the candidate genes involved in the biologic pathway of OSA. The whole genome scan identified chromosomes 2p 及19p and chromosomes 8q was associated with AHI in Caucasian and African American, respectively, which is independent of BMI. Also, the whole genome SNP array identified candidate genes associated with OSA as C-reactive protein (C-RP) and glial cell line-derived neurotrophic factor (GDNF) in European Americans and rs9526240 within serotonin receptor 2a (HTR2A) in African Americans. We identified 37 candidate genes involved in six biologic pathways of OSA including oxidative phosphorylation, cell signaling, apoptosis, cellular adhesion and motility, cell cycle, and cytokine/chemokine. Furthermore, three models were constructed to predict the sequel and response to 4-week and 12-week CPAP treatment, respectively.

Since the presentations of OSA are different among races, hence database of Taiwanese patients with OSA is urgently needed to clarify molecular mechanisms. Through recruiting the patients of moderate-severe OSA (index proband) and their first and second-degree family members, and friends and their family members (control family) and via candidate genes reported in the literature and whole genome SNP array, this project aims to achieves following goals (1) Investigating the phenotyping and familial aggregation of OSA (2) Investigating the association of genotyping on phenotyping of OSA (3) Investigating the candidate genes and the involved biologic pathways of OSA. The anticipated contributions of the results include (1) Highlighting the promise of patient-tailored management (2) Establishing an invaluable database of phenotyping and genotyping of OSA for future research (3) Promoting production of biotechnology patent and business.

ELIGIBILITY:
Inclusion Criteria:

* all participants needing age > 20 y/o
* Index proband: OSA diagnosed by overnight polysomnography (AHI>30 or AHI>15 needing therapeutic intervention)
* Index family: first-degree, second-degree relatives, or spouse of index proband
* Control proband: friends recommended by index proband, who lived in the same environment as index proband
* Control family: first-degree, second-degree relatives, or spouse of control proband

Exclusion Criteria:

* Severe CHF, COPD, CKD
* Psychiatric disorder who can't coordinate to receive evaluation
* Autoimmune disorders
* Other sleep disorders
* Refusing to anticipate or involving other study at the same time

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: moderate to severe OSA from primary care clinic friends and families from recommendation of OSA patients
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Family aggregation of OSA and its phenotype | within the first half year after enrollment
  Phenotypes assessment by PSG, craniofacial image, Hypercapnic ventilatory response testing, psychomotor vigilance task, MSLT, blood biochemistry testing, abdominal MRI, and 24 hr ambulatory BP monitor Family aggregation assessed by family-based study design (1. to compare risk of OSA between index and control proband; 2. to compare risk between index proband with more than one families suffering OSA and without; 3. to calculate inter-generation and intra-generation association index of AHI)
Association between phenotype and genotype of OSA | within the first half year after enrollment
  Genotypes assessed by candidate genes identification or whole genome SNP array Phenotypes assessment by PSG, craniofacial image, Hypercapnic ventilatory response testing, psychomotor vigilance task, MSLT, blood biochemistry testing, abdominal MRI, and 24 hr ambulatory BP monitor Association assessed by linkage study and association study

CONTACTS AND LOCATIONS:
Overall Officials: Peilin Lee, M.D, Ph.D., Principal Investigator — Center of sleep disorders, National Taiwan University Hospital
Locations (1):
- Center of sleep disorders, National Taiwan University Hospital, Taipei, Taiwan